CLINICAL TRIAL: NCT00147303
Title: Effect of Sarpogrelate on Platelet Aggregation in Patients With Cerebral Infarction: Clinical-pharmacological Dose-response Study.
Brief Title: Effect of Sarpogrelate on Platelet Aggregation in Patients With Cerebral Infarction: Dose-responsive Clinical Pharmacology Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: General Manager, Clinical Research Department I, Mitsubishi Tanabe Pharma Corporation
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI9042-17
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — sarpogrelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group L (Experimental): 25mg sarpogrelate
  Interventions: Drug: MCI-9042
- group M (Experimental): 50mg sarpogrelate
  Interventions: Drug: MCI-9042
- group H (Experimental): 100mg sarpogrelate
  Interventions: Drug: MCI-9042

INTERVENTIONS:
Drug: MCI-9042

SUMMARY:
Sarpogrelate is an antiplatelet agent that decreases 5-hydroxytryptamine( 5-HT )levels in platelets via blockade of 5-HT2 receptors, has been used in atherosclerotic peripheral arterial disease.

The present double-blind controlled clinical pharmacology study was performed on 45 patients with cerebral infarction, who were given 75, 150, or 300 mg three times daily of sarpogrelate for 7 days in order to evaluate the dose-response relationship in terms of the precisely measured inhibition of platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral infarction except cardiac source of embolism based on the NINDSⅢclassification
2. Neurological signs persisting≧ 1 day from onset
3. Defined onset of symptoms, and stable condition at the period of enrollment
4. CT or MRI detection of responsible site
5. age≧20
6. Systolic pressure≦180 mmHg, Diastolic pressure≦110 mmHg
7. The maximum intensity of platelet aggregation is above 15 % induced by serotonin (1µM) and epinephrine (3µM) on the day of prior to the first medication
8. Written informed consent must be obtained from the patients before enrollment into the study

Exclusion Criteria:

1. Functional outcome at randomization: Modified Rankin Scale=4, 5
2. Previous or planned for vascular surgery to cerebral infarction
3. History of intracranial hemorrhage
4. History of systemic bleeding, or other history of bleeding diathesis or coagulopathy
5. With severe complications ( renal or hepatic insufficiency, heart failure, hemopathy, and so on )
6. Treating malignant tumor
7. Pregnant or possibly pregnant women, or nursing mothers
8. History of sarpogrelate sensitivity
9. Previously entered in other clinical trials within 3 months
10. Less than 3 months since any other clinical trial
11. Judged by investigator to be unsuitable for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The maximum intensity of platelet aggregation on the last day of medication and as post-treatment percentage inhibition of the maximum intensity of platelet aggregation at baseline [(baseline - post-treatment )/baseline × 100 in each subject].

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Uchiyama, MD, Study Chair — Tokyo Women's Medical University

REFERENCES:
- [Result] Uchiyama S, Ozaki Y, Satoh K, Kondo K, Nishimaru K. Effect of sarpogrelate, a 5-HT(2A) antagonist, on platelet aggregation in patients with ischemic stroke: clinical-pharmacological dose-response study. Cerebrovasc Dis. 2007;24(2-3):264-70. doi: 10.1159/000105135. Epub 2007 Jul 4. PMID 17622759